CLINICAL TRIAL: NCT06648174
Title: The Project for Managing Cardiometabolic Risk in Women Diagnosed With Gestational Diabetes Mellitus: The Development and Application of "a Lifestyle Intervention Based on Health Belief Model Supported by Mobile Health"
Brief Title: The Project for Managing Cardiometabolic Risk in Women Diagnosed With Gestational Diabetes Mellitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202403080RIND
Record Dates: First submitted 2024-09-18; First posted 2024-10-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Gestational Diabetes Mellitus; Continuous Glucose Monitoring
Keywords: Gestational Diabetes Mellitus; Continuous Glucose Monitoring; Health Interventions
MeSH Terms: conditions — Diabetes, Gestational | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Controlled group-Blood glucose meters (BGM) group (Other): The participants will receive structured questionnaires at 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, and 4-12 weeks postpartum, respectively.
  Participants are required to use blood glucose meters (BGM) at "24-32 weeks of pregnancy" and "33 weeks to before delivery". After 7-14 days of glucose monitoring at "24-32 weeks of pregnancy", glucose monitor reports will be given to the participants. After the 7-14 days of glucose monitoring at "33 weeks to before delivery ", another glucose monitor reports will be given to the participants.
  Interventions: Other: Blood glucose meters (BGM)
- Experimental group1-Continuous glucose monitoring (CGM) group (Experimental): The participants will receive structured questionnaires at 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, and 4-12 weeks postpartum, respectively.
  Participants will receive a set of continuous glucose monitor (CGM) respectively at "24-32 weeks of pregnancy (first set)" and "33 weeks of pregnancy to before delivery (second set)". After 7-14 days of glucose monitoring at "24-32 weeks of pregnancy", glucose monitor reports will be given to the participants. After the 7-14 days of glucose monitoring at "33 weeks to before delivery ", another glucose monitor reports will be given to the participants.
  Interventions: Device: Continuous glucose monitor
- Experimental group2-Continuous glucose monitoring (CGM) with nursing care group (Experimental): The participants will receive structured questionnaires at 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, and 4-12 weeks postpartum, respectively.
  Participants will receive a set of continuous glucose monitor (CGM) respectively at "24-32 weeks of pregnancy (first set)" and "33 weeks of pregnancy to before delivery (second set)". After 7-14 days of glucose monitoring at "24-32 weeks of pregnancy", glucose monitor reports will be given to the participants. After the 7-14 days of glucose monitoring at "33 weeks to before delivery ", another glucose monitor reports will be given to the participants.
  Participants will receive nursing care for gestational diabetes at 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, and 4-12 weeks postpartum.
  Interventions: Device: Continuous glucose monitor; Behavioral: Perinatal nursing care for gestational diabetes

INTERVENTIONS:
Device: Continuous glucose monitor — Participants will receive a set of continuous glucose monitor (CGM) at 24-32 weeks of pregnancy (first set); and 33 weeks of pregnancy to before delivery (second set) respectively.
  CGM wearing instruction will be provided before the first wearing at 24-32 weeks of pregnancy. After completing the first wearing (approximately 7-14 days after starting to wear), the investigators will provide glucose monitor reports. The second CGM was worn from the 33rd week of pregnancy to before delivery, and another glucose monitor reports was given approximately 7-14 days after starting to wear.
  Other Names: Abbott FreeStyle Libre 2 (CGM)
  Arms: Experimental group1-Continuous glucose monitoring (CGM) group; Experimental group2-Continuous glucose monitoring (CGM) with nursing care group
Behavioral: Perinatal nursing care for gestational diabetes — Individual nursing care and consultation for women with gestational diabetes mellitus, including glucose monitor suggestions, dietary suggestions, emotional support, breastfeeding support at 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, and 4-12 weeks postpartum.
  Arms: Experimental group2-Continuous glucose monitoring (CGM) with nursing care group
Other: Blood glucose meters (BGM) — Participants are required to use blood glucose meters (BGM) at 24-32 weeks of pregnancy and 33 weeks to before delivery. After 7-14 days of glucose monitoring at 24-32 weeks of pregnancy, glucose monitor reports will be given to the participants. After the 7-14 days of glucose monitoring at 33 weeks to before delivery, another glucose monitor reports will be given to the participants.
  Arms: Controlled group-Blood glucose meters (BGM) group

SUMMARY:
This study aims to examine the effects of a lifestyle intervention based on a health belief model (HBM) supported by mobile health (mHealth) and the impact of continuous glucose monitoring (CGM) on maternal glycemic parameters, cardiometabolic risk, health behavior and infant's outcomes among women diagnosed with gestational diabetes mellitus (GDM).

DETAILED DESCRIPTION:
Background: Women with gestational diabetes mellitus (GDM) are more likely to develop cardiometabolic risk (CMR). CMR refers to the risk factors that promote the chance of developing type 2 diabetes mellitus or cardiovascular events. However, using a family-centered approach, the effectiveness of continuous administration of both mobile health management and theoretical based lifestyle intervention from pregnancy to postpartum in preventing women at high risk of GDM from developing CMR has rarely been studied.

Methods: This randomized controlled trial will recruit 120 GDM pregnant women in northern Taiwan. The participants will be randomly assigned to the control group (blood glucose meters (BGM); n=40 people), intervention group 1 (continuous glucose monitoring (CGM); n=40 people), intervention group 2 (HBM-based lifestyle and mHealth intervention + CGM; n=40 people).The comparison group will receive the routine care and finger-prick test for blood glucose monitoring (BGM) during pregnancy.The intervention group 1 will receive CGM during pregnancy. The intervention group 2 will receive a HBM-based lifestyle and mHealth management program on 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery, 4-12 weeks postpartum, including CGM during pregnancy.We intend to compare outcome variables among three groups. The outcomes variables will be assessed at baseline (24-32 weeks of pregnancy), 33 weeks of pregnancy to before delivery, 4 to 12 weeks after delivery. The primary outcomes were maternal glycemic parameters, cardiometabolic risk factors, and maternal health behavior. Outcomes will be assessed at baseline (24-32 weeks of pregnancy), 33 weeks of pregnancy to before delivery, 4 to 12 weeks after delivery. Generalized estimating equation (GEE) will be used to examine the trajectories and the effectiveness of the project for managing cardiometabolic risk on cardiometabolic risk and health behavior.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or above
2. Pregnant women diagnosed with gestational diabetes mellitus
3. Willing to participate in the study

Exclusion Criteria:

1. Diagnosed with diabetes mellitus before pregnancy
2. Allergic to materials such as tapes (e.g., redness, swelling, itching, pain, blisters, or rashes caused by breathable tapes or patches)
3. Abnormal coagulation function

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The participants of this study are pregnant women with gestational diabetes mellitus.
Enrollment: 120 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Abnormal Maternal Oral Glucose Tolerance Test Results | 24-32 weeks of pregnancy, 4-12 weeks postpartum
  This outcome measure assesses the number of participants with abnormal results from the Oral Glucose Tolerance Test (OGTT), which includes measurements of fasting, 1-hour, and 2-hour glucose levels. The data will be summarized based on the thresholds established for abnormal glucose levels, as per standard diagnostic criteria for gestational diabetes.
HOMA-IR Value for Assessing Insulin Resistance in Participants | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery and 4-12 weeks postpartum
  This outcome measure evaluates the HOMA-IR (Homeostasis Model Assessment of Insulin Resistance) value in participants, calculated using fasting insulin and fasting glucose levels. Data will be obtained through reviews of medical records.
Total Cholesterol Levels in Participants | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery and 4-12 weeks postpartum
  This outcome measure assesses the total cholesterol levels in participants. Data will be obtained through reviews of medical records. The data will be summarized by reporting the mean total cholesterol level, as well as the proportion of participants classified as having high total cholesterol levels based on established clinical thresholds.
Triglycerides Levels in Participants | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery and 4-12 weeks postpartum
  This outcome measure assesses the triglycerides levels in participants. The data obtained through medical record reviews. The data will be summarized by reporting the mean triglycerides level, as well as the proportion of participants classified as having high triglycerides levels based on established clinical thresholds.
High-density Lipoprotein Levels in Participants | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery and 4-12 weeks postpartum
  This outcome measure assesses the high-density lipoprotein levels in participants. The data obtained through medical record reviews. The data will be summarized by reporting the mean high-density lipoprotein level, as well as the proportion of participants classified as having high high-density lipoprotein levels based on established clinical thresholds.
Low-density Lipoprotein Levels in Participants | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery and 4-12 weeks postpartum
  This outcome measure assesses the low-density lipoprotein levels in participants. The data obtained through medical record reviews. The data will be summarized by reporting the mean low-density lipoprotein level, as well as the proportion of participants classified as having high low-density lipoprotein levels based on established clinical thresholds.
Glycated Albumin Levels in Participants | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery and 4-12 weeks postpartum
  This outcome measure assesses the glycated albumin levels in participants. The data obtained through medical record reviews. The data will be summarized by reporting the mean glycated albumin level, as well as the proportion of participants classified as having high glycated albumin levels based on established clinical thresholds.
Fasting Plasma Glucose Levels in Participants | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery and 4-12 weeks postpartum
  This outcome measure assesses the fasting plasma glucose levels in participants. The data obtained through medical record reviews. The data will be summarized by reporting the mean fasting plasma glucose level, as well as the proportion of participants classified as having high fasting plasma glucose levels based on established clinical thresholds.
Incidence of Fetal Macrosomia as Measured by Birth Weight | 4-12 weeks postpartum
  This outcome measure assesses the incidence of fetal macrosomia in participants. Data will be summarized by reporting the proportion of newborns classified as having fetal macrosomia based on the established weight threshold.

SECONDARY OUTCOMES:
Incidence of Hypertensive Disorders in Pregnancy | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery
  This outcome measure assesses the incidence of hypertensive disorders in pregnancy, including gestational hypertension, preeclampsia, and eclampsia. Data will be summarized by reporting the proportion of participants diagnosed with any hypertensive disorder during pregnancy.
Rate of Cesarean Section Deliveries | 4-12 weeks postpartum
  This outcome measure assesses the rate of cesarean section deliveries among participants.
Health Belief Scale for Glycemic Control | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery
  A 21-item Likert scale based on the Health Belief model includes 5 categories: perceived susceptibility, perceived severity, perceived benefits, perceived barriers and self-efficacy.
Glucose monitoring satisfaction Scale | 33 weeks of pregnancy to before delivery
  Satisfaction of using continuous glucose monitoring (CGM) or blood glucose meters (BGM) access by Likert scale. A 4-item Likert scale includes 4 categories: ease of use, painful, convenience and overall satisfaction. Each item scores from 1-5. A higher score means lower satisfaction.
Perceived benefits and barriers of CGM assessed by Benefits of CGM (BenCGM) and Burdens of CGM (BurCGM) Questionnaires | 33 weeks of pregnancy to before delivery
  The Benefits of Continuous Glucose Monitoring (BenCGM) and Burdens of Continuous Glucose Monitoring (BurCGM) Questionnaires will be used to assess participants' perceived benefits and barriers of using CGM. The data will be summarized as quantitative scores, with higher scores indicating greater perceived benefits or barriers, respectively. Each questionnaire includes multiple items rated on a Likert scale, and the total scores will be aggregated for each participant.
Gestational Weight Gain as Measured by Weight Change Across Pregnancy Weeks or Total Weight Gain During Pregnancy | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery
  This outcome measure assesses gestational weight gain in participants, defined as the weight change between different pregnancy weeks or the total weight gain during pregnancy.
Depression Severity as Measured by the Edinburgh Postnatal Depression Scale (EPDS) | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery and 4-12 weeks postpartum
  This outcome measure assesses the severity of depression in participants using the Edinburgh Postnatal Depression Scale (EPDS), a 10-item questionnaire. Each item is scored from 0 to 3, resulting in a total score range from 0 to 30. Higher scores indicate a higher likelihood of depression, with scores above 12 or 13 suggesting probable depression.
Infant Growth Curve as Measured by WHO Growth Standards | 4-12 weeks postpartum
  This outcome measure assesses infant growth curves using the World Health Organization (WHO) growth standards. Data on infant weight, length, and head circumference will be collected at multiple time points. The data will be summarized by reporting the mean values at each time point and the proportion of infants classified as underweight, normal weight, or overweight.
Average Postpartum Weight Retention | 24-32 weeks of pregnancy, 4-12 weeks postpartum
  The postpartum weight retention will be measured as the difference between pre-pregnancy weight and weight at 4-12 weeks postpartum
Percentage of Participants on Insulin Medications | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery and 4-12 weeks postpartum
  This outcome will report the proportion of participants who required insulin medications, expressed as a percentage of the total study population. Insulin use will be tracked through medical records and self-reports.
Average Exercise Frequency | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery and 4-12 weeks postpartum
  Exercise frequency will be measured based on self-reported exercise sessions per week. The data will be summarized as an average number of sessions per week for the study population at each time point.
Health behavior change of glycemic control Scale | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery and 4-12 weeks postpartum
  A 3-item Likert scale based on the Transtheoretical model, including self-monitoring of glucose level, diet and physical activity. Each item scores from 0-4. A higher score means closer to the action or maintenance stage.
Assessment of Quality of Life Using the World Health Organization Quality of Life Scale (WHOQOL-BREF) Taiwan Version | 24-32 weeks of pregnancy, 33 weeks of pregnancy to before delivery and 4-12 weeks postpartum
  This measure assesses quality of life using the WHOQOL-BREF Taiwan version. Data will be aggregated and reported as domain-specific scores and an overall quality of life score, based on participant responses.

CONTACTS AND LOCATIONS:
Overall Officials: HUNG-HUI CHEN, PhD, Principal Investigator — National Taiwan University Hostiptal
Locations (1):
- National Taiwan University Hospital Hsin-Chu Branch BioMedical Park Hospital, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No